CLINICAL TRIAL: NCT06527326
Title: the Study of the Association Between the Gut Microbiota and Central Serous Chorioretinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-0611
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Central Serous Chorioretinopathy
Keywords: central serous chorioretinopathy; Bifidobacterium genus; the gut dysbiosis
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receiving Bifidobacterium supplements (Experimental)
  Interventions: Dietary Supplement: Live Combined Bifidobacterium
- receiving placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Live Combined Bifidobacterium — the Bifidobacterium genus supplement
  Arms: receiving Bifidobacterium supplements
Dietary Supplement: Placebo — Placebo
  Arms: receiving placebo

SUMMARY:
To investigate the potential association between gut microbiota and central serous chorioretinopathy (CSC), we have observed in our clinical practice that CSC patients often experience chronic gastrointestinal issues. This observation has led us to hypothesize that CSC may be associated with gut dysbiosis. The Bifidobacterium genus is widely recognized as a beneficial gut bacterium, and numerous well-established Bifidobacterium supplements are available on the market. To explore this possible connection, we will collect fecal samples from both CSC patients and healthy individuals. Using whole-metagenome shotgun sequencing, we will compare the gut microbiota compositions of the two groups to determine if significant differences exist. Additionally, we will randomly assign patients to two groups: one group will receive Bifidobacterium supplements for at least one month, while the other group will receive a placebo. We will then assess whether the group receiving the supplements experiences faster recovery and lower relapse rates compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Diagnosis of acute central serous chorioretinopathy (CSC) (affected eye: ① FFA and ICGA showing typical CSC manifestations, ② presence of subretinal fluid (SRF) at the macular fovea, ③ disease duration ≤ 6 months)
* Best Corrected Visual Acuity (BCVA): 53 to 86 letters
* Other: No significant systemic diseases, signed informed consent, and able to commit to follow-up

Exclusion Criteria:

* Presence of significant systemic diseases
* BCVA of 20/200 or worse
* Presence of choroidal or retinal atrophy in the macular fovea of the affected eye
* Presence of choroidal neovascularization (CNV), age-related macular degeneration (AMD), polypoidal choroidal vasculopathy (PCV), diabetic retinopathy (DR), choroidal hemangioma, pigment epithelial detachment (PED), etc., in the affected eye
* High myopia in the affected eye

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | through study completion, an average of one year
  BCVA is commonly assessed during eye exams to determine the effectiveness of vision correction and to evaluate the impact of eye conditions or diseases on vision.

SECONDARY OUTCOMES:
Central Retinal Thickness (CRT) | through study completion, an average of one year
  Central Retinal Thickness is typically assessed using imaging techniques such as optical coherence tomography (OCT), which provides detailed cross-sectional images of the retina, allowing for accurate measurement of its thickness.
the thickness of Subretinal Fluid (SRF) | through study completion, an average of one year
  Subretinal fluid can cause vision distortion and may require medical intervention to address the underlying condition and reduce fluid accumulation.
the thickness of Choroid | through study completion, an average of one year
  Choroidal hyperpermeability is one of the key mechanisms underlying the pathogenesis of central serous chorioretinopathy (CSC).
Choroidal Vascular Index (CVI) | through study completion, an average of one year
  This is a ratio or index that quantifies the proportion of the choroid occupied by blood vessels compared to the total choroidal area. It provides a measure of the relative density of the choroidal vasculature.
Choroidal Vascular Volume (CVV) | through study completion, an average of one year
  This measures the total volume of the choroidal blood vessels within a specific area of the choroid. It reflects the overall blood vessel density and the amount of blood flowing through the choroidal vasculature.

CONTACTS AND LOCATIONS:
Overall Officials: Panpan Ye, doctor, Principal Investigator — 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejiang, China